CLINICAL TRIAL: NCT06146608
Title: Heme and Non-heme Iron Intakes, Gut Microbiota, and Influence on Host Iron Absorption
Acronym: FeMicrobiome
Status: Recruiting | Type: Observational
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB0147198; 2023-67017-39059 (Other Grant/Funding Number: United States Department of Agriculture)
Record Dates: First submitted 2023-07-11; First posted 2023-11-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Anemia, Iron Deficiency; Iron Overload
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma samples and fecal DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The FeMicrobiome study will evaluate gut microbiome features and their relationships with dietary iron absorption in healthy adults. The investigators hypothesize that (1) the gut microbiota can be shaped by the heme and non-heme Fe content of the diet and that (2) this will influence individual variation in dietary Fe absorption.

DETAILED DESCRIPTION:
Iron is an essential micronutrient ingested as either heme iron (from animal products) or non-heme iron (from both plant and animal sources). Humans have no regulatable means of eliminating absorbed iron, necessitating tight control of dietary iron absorption. Likewise, native microbes have evolved efficient iron sensing and utilization pathways to scavenge iron from the gastrointestinal environment, resulting in a competition for iron between the host and their microbiota. As growing numbers of Americans adopt plant-based diets, heme iron intakes are markedly reduced. This may shift the gut microbiome as some gut microbiota cannot independently synthesize heme and require host dietary heme sources to support their heme-dependent functions. Animal data have recently discovered that other gut microbiota respond to a low iron. To date, significant knowledge gaps exist on the interplay between dietary iron sources, native gut microbes, and iron utilization in humans. In the FeMicrobiome study, study investigators will recruit 120 adults who habitually ingest plant-based diets or habitually ingest diets containing animal protein (e.g., beef, pork, chicken, fish, and seafood). Iron absorption will be measured by using an in vivo, functional approach based on stable iron isotopes (i.e., 57Fe). Study participants will consume 57Fe (as ferrous sulfate) in the fasted state followed by two standardized meals. Two weeks after iron dosing, a blood sample will be collected from each participant and the amount of 57Fe incorporated into red blood cells will be measured using magnetic sector thermal ionization mass spectrometry. A stool sample will be collected near the time of 57Fe consumption. DNA will be extracted from this stool sample and sequenced using a high-depth shotgun metagenomic approach.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Age between 18- 40y
* Non-smoking
* Not currently taking vitamin, mineral, prebiotic, and probiotic supplements.
* Females: premenopausal and not pregnant or lactating
* No preexisting medical complications (such as eating disorders, hemoglobinopathies, malabsorption diseases, steroid use, substance abuse history, or taking medications known to influence iron homeostasis)
* Body mass index (BMI) between 18 - 27 kg/m2.

Exclusion Criteria:

* BMI <18 or > 27 kg/m2,
* Age <18 y or > 40y,
* Smoking
* Pregnancy, lactating
* Have gastrointestinal disorders/malabsorption diseases/hemoglobinopathies/dietary restrictions/steroid use/ medication use of medications known to impact iron status, iron utilization or inflammatory status
* Currently take vitamin, mineral, prebiotic, and probiotic supplements.
* Recently received antibiotic treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 120 healthy adults who habitually consume plant-based diets or habitually consume diets containing animal protein
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
The percent of non-heme iron absorption | 2-week
  Percent non-heme iron absorption will be determined by red blood cell iron incorporation of stable 57Fe
The concentrations of hemoglobin | baseline
  The concentrations of hemoglobin (d/dL)
The concentrations of ferritin | baseline
  The concentrations of ferritin (ug/L)
Serum transferrin receptor | baseline
  Serum transferrin receptor in mg/L
The hematocrit | baseline
  Blood hematocrit in %
Habitual dietary information | baseline
  Habitual dietary information will be obtained from Diet History Questionnaire III.
Dietary information on the day prior to iron dosing | baseline
  Detailed dietary information about all foods and beverages consumed on the day prior to iron dosing will be obtained from the Automated Self-Administered 24-Hour Dietary Assessment Tool. Total iron intake will be presented as a proportion of the daily iron requirement. Total heme and non-heme iron intakes will be quantified.
Gut microbiome composition | baseline
  Shotgun metagenomic sequencing will be performed to assess the gut microbiome compositions and gene functional features in a stool sample collected within one day before or after iron dosing.

CONTACTS AND LOCATIONS:
Overall Officials: KIMBERLY ORA OBRIEN, PhD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided